CLINICAL TRIAL: NCT00038298
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose Ranging Study to Assess the Efficacy, Safety and Tolerability of AMG 719 in Subjects With Rheumatoid Arthritis Receiving Methothrexate
Brief Title: A Rheumatoid Arthritis (RA) Study Treating Signs and Symptoms of RA in People With RA & Receiving Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20010238
Record Dates: First submitted 2002-05-29; First posted 2002-05-31 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 50 mg (Experimental): 50 mg 3 times weekly
  Interventions: Drug: AMG 719
- 400 mg (Experimental): 400 mg 3 times weekly
  Interventions: Drug: AMG 719
- 200 mg (Experimental): 200 mg 3 times weekly
  Interventions: Drug: AGM 719
- Placebo (Placebo Comparator): Placebo comparator associated with each active arm. (3:1 active vs placebo)
  Interventions: Drug: Placebo; Drug: placebo to AMG 719

INTERVENTIONS:
Drug: Placebo — Placebo given 3 times weekly
  Arms: Placebo
Drug: AMG 719 — 50 mg 3 times weekly
  Arms: 50 mg
Drug: AGM 719 — 200 mg 3 times weekly
  Arms: 200 mg
Drug: AMG 719 — 400 mg 3 times weekly
  Arms: 400 mg
Drug: placebo to AMG 719 — Placebo dose given 3 times weekly
  Arms: Placebo

SUMMARY:
This clinical study is investigating AMG 719, an investigational drug, for the treatment of patients who have Rheumatoid Arthritis and who are taking Methotrexate. AMG 719 is a drug which is self-injected beneath the skin (similarly to the way insulin is self-injected by diabetics). Patients on this study are on study for 28-weeks. They visit the study facility at least 11 times while participating in the study.

ELIGIBILITY:
* Men or women, at least 18 years of age at screening
* Diagnosed with Rheumatoid Arthritis, with a disease duration of at least 24 weeks, receiving methotrexate, and having no recent history of substance or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2002-04; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
AMG 719 has a favorable safety profile in subjects with RA receiving methotrexate. | Week 24

SECONDARY OUTCOMES:
To assess the effects of multiple doses of AMG 719 relative to placebo on signs and symptoms of RA | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_47_AMG_719_20010238.pdf